CLINICAL TRIAL: NCT03622944
Title: Servikal bölge Patolojisi Olan Bireylerde Egzersiz ve Manuel Terapi yöntemlerinin ağrı, postür ve yaşam Kalitesi üzerindeki etkinliğinin Belirlenmesi
Brief Title: Effect of Exercise and Manuel Therapy Methods on Pain, Posture, Daily Living in People With Cervical Pathologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO15/564
Record Dates: First submitted 2018-07-18; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Musculoskeletal Disorder of the Neck
Keywords: neck pain; physiotherapy; rehabilitation
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Muscle energy technic (Active Comparator): post isometric relaxation technics were used as muscle energy technics.
  Interventions: Procedure: Muscle Energy Technic; Procedure: Exercise
- Deep Friction Massage (Active Comparator): Painful areas palpated and deep friction massage was applied.
  Interventions: Procedure: Deep Friction Massage; Procedure: Exercise
- exercise (Active Comparator): Physiotherapist guided Spinal stabilization exercises were applied.
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Muscle Energy Technic — post isometric relaxation technics were applied to levator scapulae, trapezius, pectoralis muscles three sessions per week, totally six weeks.
  Arms: Muscle energy technic
Procedure: Deep Friction Massage — deep friction massage was applied to cervical region included tendons, muscles and soft tissue.
  Arms: Deep Friction Massage
Procedure: Exercise — spinal stabilization exercise were applied three sessions in a week totally six weeks.

SUMMARY:
The aim of the study is to determine the effect of exercise and two different manual therapy methods on pain, quality of life and posture in people with neck pain.

DETAILED DESCRIPTION:
Deep friction massage will use on cervical regions in first group, muscle energy technic will use second group and cervical stabilization exercise will use as an third group. For all groups, pain intensity, Quality of life and posture will assess.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of cervical disorder (for example; chronic neck pain, cervical disc herniation)
* must have pain at least three months.

Exclusion Criteria:

* History of structural scoliosis
* History of surgery
* History of metabolic, neurologic and metastatic diseases.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
change in pain sensitivity | change from baseline PPT at six weeks
  pressure pain threshold (PPT) was measured with digital algometer. Pressure pain threshold which identifies minimum levels increasing mechanical stimulus is gold standard method for measuring pain sensitivity. PPT was measured from cervical vertebrae's spinous process and muscle belly's. Algometer range was set 0 kgF to 12kgF. Higher values represent increased pressure sensation.

SECONDARY OUTCOMES:
change in Light touch sensation | change from baseline light touch sensation at six weeks
  Semmes weinstein monofilaments were used to determine light touch sensation. It has twenty different evaluator size. Evaluator size was started 2.83 point and higher values represent worse outcome. Upper extremity dermatomes were tested.
change in upper extremity disability | Change from baseline disability at six weeks .
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire was used.The questionnaire has 34 item which each item scored 1 to 5 points. All responses summed and averaged.This value is then transformed to a score out of 100 by subtracting one and multiplying by 25. This transformation is done to make the score easier to compare to other measures scaled on a 100 scale. Minimum score is "0" and total score is "100". higher values represent a worse outcome.
change in posture | change from baseline posture at six weeks
  Posture was assessed with global postural system. This computer generated system has two cameras and lets three different plane postural assessment. the assessments and postural deviation calculate with computer programme.
change in perceived life quality | change from baseline life quality at six weeks
  perceived quality of life was assessed with nottingham health profile. the questionnaire has 38 questions in 6 subareas, with each question assigned a weighted value; the sum of all weighted values in a given subarea adds up to 100. higher values represent better life quality.
change in functional disability | change from baseline functional disability at six weeks
  Neck Disability Index (NDI) was used.NDI total scores ranged from 0 (no disability) to 50 (severe disability) which have ten items assessing perceived neck pain during daily living activities such as lifting, reading, driving, sleeping and recreational activities.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, PhD, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rihn JA, Radcliff K, Hipp J, Vaccaro AR, Hilibrand AS, Anderson DG, Albert TJ. Radiographic variables that may predict clinical outcomes in cervical disk replacement surgery. J Spinal Disord Tech. 2015 Apr;28(3):106-13. doi: 10.1097/BSD.0b013e31826a0c84. PMID 24694684
- [Result] Carreon LY, Glassman SD, Campbell MJ, Anderson PA. Neck Disability Index, short form-36 physical component summary, and pain scales for neck and arm pain: the minimum clinically important difference and substantial clinical benefit after cervical spine fusion. Spine J. 2010 Jun;10(6):469-74. doi: 10.1016/j.spinee.2010.02.007. Epub 2010 Apr 1. PMID 20359958
- [Result] Persson LC, Lilja A. Pain, coping, emotional state and physical function in patients with chronic radicular neck pain. A comparison between patients treated with surgery, physiotherapy or neck collar--a blinded, prospective randomized study. Disabil Rehabil. 2001 May 20;23(8):325-35. doi: 10.1080/09638280010005567. PMID 11374522
- [Result] Boyles R, Toy P, Mellon J Jr, Hayes M, Hammer B. Effectiveness of manual physical therapy in the treatment of cervical radiculopathy: a systematic review. J Man Manip Ther. 2011 Aug;19(3):135-42. doi: 10.1179/2042618611Y.0000000011. PMID 22851876